CLINICAL TRIAL: NCT05761080
Title: Fast Track Therapeutic Model in Acute Complicated Appendicitis in Pediatrics
Acronym: FTAA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-FAS-2020-120
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Appendectomy; Complicated Appendicitis; Periappendicular Abscess
Keywords: Complicated appendicitis
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental branch (Experimental): Patients will be included in the study during the anesthetic surgery evaluation.
  The patient will be randomized at the time of informed consent to know the postoperative guideline to be used.
  Randomization of patients on postoperative day 3.
  If patient belong to the Fast Track group:
  Application of discharge criteria in the experimental branch at 72 hours post-surgery, and administration of oral antibiotic therapy: Amoxicillin - clavulanic acid, dose: 100mg/Kg/day every 8 hours for a total of 5 days.
  There will be a follow-up at 5, 7 and 30 days after discharge. In addition, there will be a face-to-face visit 2 weeks after the intervention.
  Interventions: Drug: Amoxicillin clavulanic acid IV 3 days and PO until day 5
- Control branch (Active Comparator): Patients will be included in the study during the anesthetic surgery evaluation.
  The patient will be randomized at the time of informed consent to know the postoperative guideline to be used.
  Randomization of patients on postoperative day 3.
  If patient belongs to the control group:
  Application of discharge criteria in control branch 5 days postoperative, according to current clinic guidelines. Administration of Amoxicillin - clavulanic acid, dose: 100mg/Kg/day every 8 hours, intravenous during 5 days
  There will be a follow-up at 5, 7 and 30 days after discharge. In addition, there will be a face-to-face visit 2 weeks after the intervention.
  Interventions: Drug: Amoxicillin clavulanic acid IV during hospitalization

INTERVENTIONS:
Drug: Amoxicillin clavulanic acid IV during hospitalization — Amoxicillin clavulanic acid IV 5 days during hospitalization. Application of discharge criteria at 5 postoperative days, according to guidelines current clinic.
  Arms: Control branch
Drug: Amoxicillin clavulanic acid IV 3 days and PO until day 5 — Amoxicillin clavulanic acid IV 3 days during hospitalization and at discharge Amoxicillin clavulanic acid PO until day 5.
  Application of discharge criteria at 72 postoperative hours, administering oral antibiotic therapy with a spectrum similar to that of the control group total of 5 days and sending the patient home with oral analgesia.
  Arms: Experimental branch

SUMMARY:
Evaluate the application of the new therapeutic model post Fast Track surgery, in complicated acute appendicitis, in pediatric population on the rate of complications postoperative in the form of abdominal abscesses.

DETAILED DESCRIPTION:
Complicated appendicitis is defined as the finding in the intraoperative study of a perforated, gangrenous or contaminated appendix with the presence of periappendicular abscess. In November 2005, the synthesis of an "Evidence-based clinical practice guide for acute appendicitis in pediatrics" at the Hospital Vall d'Hebron, the result of a committee of experts in the field. This protocol has been the guideline for our center in recent years.

Currently, the therapeutic approach is based on monotherapy antibiotic management (except for drug allergies, appendicular peritonitis, immunosuppression or nosocomial acquisition) in the postoperative period, with a minimum duration of 5 days (intravenous treatment). Therefore, the minimum hospital stay in these patients is expected to be equal to or more than 5 days.

Acute appendicitis represents the most frequent cause of acute abdomen in pediatric patients older than two years. It affects approximately 80,000 children in the European Union, making appendectomy one of the most frequent non-elective pediatric interventions performed by pediatric surgeons.

In recent years, several ambispective studies have been carried out at national level applying new therapeutic models that allow shortening the hospital stay by applying more lax discharge criteria and reducing the duration of intravenous antibiotic treatment, without significant alterations in the rate of postoperative complications.

By reducing hospital stay, the fast-track model not only brings clinical benefits to patients, but also economic benefits to the healthcare system.

ELIGIBILITY:
Inclusion criteria:

* Ages 2 to 16 years Intraoperative diagnosis of complicated appendicitis. Laparoscopic appendectomy. 72 hours postoperative. Leukocyte count and C-reactive protein at 72 hours post-surgery increased (minimum 20% with respect to the preoperative baseline). Complete oral tolerance. Pain controlled with conventional analgesia.Afebrile (more than 24 hours).

Exclusion criteria:

* History of cystic fibrosis, Crohn's disease, transplant or appendicitis. Chronic requiring elective technique. Contraindication to the administration of amoxicillin-clavulanic acid. Refusal to participate in the study by parents/legal guardians.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication Rate | 30 days

SECONDARY OUTCOMES:
Hospital readmission rate | 30 days
Procalcitonina value | 3 days
  Blood sample
Antibiotic consumption | 30 days
Associated costs | 30 days
Quality of life measure | 30 days
  Measured by EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Martinez-Zapata, MD, PhD, Study Chair — Institut de Recerca Sant Pau
Locations (7):
- Spain (7):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Universitario Dr. Josep Trueta, Girona
  - Complejo Universitario Hospitalario de Santiago de Compostela, Santiago de Compostela
  - Hospital Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No